CLINICAL TRIAL: NCT00124943
Title: A Phase I/II Safety Trial of Intracoronary Administration of Systemic Nanoparticle Paclitaxel (ABI-007) for the Prevention of In-Stent Restenosis
Brief Title: Use of Nanoparticle Paclitaxel (ABI-007) for the Prevention of In-Stent Restenosis
Acronym: SNAPIST-III
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Responsible Party: Sponsor
Organization: Celgene (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVR003
Record Dates: First submitted 2005-07-27; First posted 2005-07-29 (Estimated); Results first posted 2012-03-08 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Coronary Restenosis
Keywords: Prevention of Instent Restenosis
MeSH Terms: conditions — Coronary Restenosis | interventions — Taxes; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 10 mg/m^2 nanoparticle paclitaxel (Experimental): Participants received a single dose of 10 mg/m^2 nanoparticle paclitaxel administered via intracoronary catheter immediately following percutaneous transluminal coronary angioplasty/stenting (de novo lesion) or balloon angioplasty (in-stent restenosis lesions).
  Interventions: Drug: Nanoparticle Paclitaxel
- 22 mg/m^2 nanoparticle paclitaxel (Experimental): Participants received a single dose of 22 mg/m^2 nanoparticle paclitaxel administered via intracoronary catheter immediately following percutaneous transluminal coronary angioplasty/stenting (de novo lesions) or balloon angioplasty (in-stent restenosis lesions).
  Interventions: Drug: Nanoparticle Paclitaxel
- 35 mg/m^2 nanoparticle paclitaxel (Experimental): Participants received a single dose of 35 mg/m^2 nanoparticle paclitaxel administered via intracoronary catheter immediately following percutaneous transluminal coronary angioplasty/stenting (de novo lesions) or balloon angioplasty (in-stent restenosis lesions).
  Interventions: Drug: Nanoparticle Paclitaxel
- 45 mg/m^2 nanoparticle paclitaxel (Experimental): Participants received a single dose of 45 mg/m^2 nanoparticle paclitaxel administered via intracoronary catheter immediately following percutaneous transluminal coronary angioplasty/stenting (de novo lesions) or balloon angioplasty (in-stent restenosis lesions).
  Interventions: Drug: Nanoparticle Paclitaxel

INTERVENTIONS:
Drug: Nanoparticle Paclitaxel — Nanoparticle albumin-bound paclitaxel, administered via intracoronary catheter.
  Other Names: ABI-007; Abraxane®; Coroxane™

SUMMARY:
The purpose of this study was to investigate the use of systemic intracoronary administration of albumin-bound paclitaxel, ABI-007, for the prevention and reduction of restenosis following de novo stenting or following angioplasty for in-stent restenosis.

DETAILED DESCRIPTION:
This study consisted of a Phase I non-randomized dose escalation phase to determine the maximum tolerated dose and a randomized Phase II component to assess preliminary efficacy. Nanoparticle paclitaxel was administered by intracoronary catheter following either successful and uncomplicated stenting of de novo lesions in native coronary arteries or following successful and uncomplicated balloon angioplasty of instent restenosis (ISR) lesions.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant and non-lactating female, and ≥ 18 years of age.
* Diagnosis of angina pectoris or unstable angina pectoris or patients with documented silent ischemia.
* Left ventricular ejection fraction ≥30%
* Patient has undergone successful and uncomplicated stenting of up to 2 de novo lesions in native coronary arteries OR patient has undergone successful and uncomplicated balloon angioplasty of up to 2 in-stent restenosis (ISR) lesions in native coronary arteries, but not both.
* Thrombolysis In Myocardial Infarction (TIMI) 3 coronary flow post-stenting for de novo lesions or post balloon angioplasty for ISR lesions.
* No angiographic evidence of thrombus post-procedure.
* Target vessel ≥2.5 mm diameter (by angiography).
* Each de novo lesion is such that it is stented with ≤ 25 mm of single continuous stent.
* Each in-stent restenosis (ISR) lesion is ≤ 25 mm in length.
* There is at least 5 mm of non-diseased vessel on either side of target lesion(s).
* By intravascular ultrasound (IVUS), stent is fully opposed and has a minimum diameter of 2.5 mm or an in-stent luminal area ≥ 5.0 mm^2
* Patient or guardian has provided a signed written informed consent to participate in the study and in all follow-up assessments using a form that is approved by the local Institutional Review Board (IRB)/Ethics Committee of the investigative site.

Exclusion Criteria:

* Target de novo lesion was treated with a drug-eluting stent
* Target ISR lesion requires any treatment other than balloon angioplasty
* Patient has both a de novo lesion and an ISR lesion.
* If more than 2 lesions are treated with percutaneous coronary intervention (PCI), or it is anticipated that additional lesions will require treatment within 2 months.
* Previous PCI within preceding two months.
* Intended surgical intervention within 6 months of enrollment in the study.
* Unprotected left main disease with >50% stenosis
* Malapposition, dissection, or unmasking of a significant narrowing in the inflow or outflow area of the implanted stent.
* Women who are pregnant and women of child bearing potential who do not use adequate contraception
* Previous participation in another study with any investigational drug or device within the past 30 days or current enrollment in any other clinical protocol or investigational drug or device trial.
* Patient has a life expectancy of less than 12 months or there are factors making clinical and/or angiographic follow-up difficult
* Any significant medical condition which, in the investigator's opinion, may interfere with the patient's optimal participation in the study
* Heart transplant candidate or recipient
* Patient is immunosuppressed or is HIV positive.
* Patient has experienced a Q wave or a non Q wave myocardial infarction (MI) with documented total creatine kinase (CK) ≥2 times normal within the preceding 24 hours and the CK and creatine kinase-MB fraction (CK-MB) enzymes remain above normal at the time of the procedure.
* Cardiogenic shock: sustained systolic blood pressure (SBP) less than 80 mmHg, with no response to fluids or SBP less than 100 mmHg with vasopressors (in absence of bradycardia)
* Any individual who may refuse a blood transfusion
* Documented major gastro-intestinal bleeding within 3 months
* The following lab values at baseline are exclusionary:

  * Serum creatinine > 2.5 mg/dl;
  * Platelet count < 150,000 cells/mm^3;
  * Absolute neutrophil count (ANC) < 2000 cells/mm^3;
  * Hemoglobin (HGB) <9 g/dl;
  * Total bilirubin >1.5 mg/dl;
  * Alanine Aminotransferase (SGPT) > 2.5 x upper limit of normal range (ULN);
  * Aspartate Aminotransferase (SGOT) > 2.5 x ULN;
  * Alkaline phosphatase > 2.5 x ULN.
* Known allergy/hypersensitivity/contraindication to the study drug; to any taxanes; or to any required study treatment: aspirin, clopidogrel bisulfate, stent materials
* Pre-existing peripheral neuropathy of National Cancer Institute (NCI) Toxicity Grade > 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2005-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose' Iglesias, MD, Study Director — Celgene Corporation

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 122 patients were randomized into the study and 112 received study medication.
Period: Phase I
Arm/Group | 10 mg/m^2 Nanoparticle Paclitaxel | 22 mg/m^2 Nanoparticle Paclitaxel | 35 mg/m^2 Nanoparticle Paclitaxel | 45 mg/m^2 Nanoparticle Paclitaxel
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Phase II
Arm/Group | 10 mg/m^2 Nanoparticle Paclitaxel | 22 mg/m^2 Nanoparticle Paclitaxel | 35 mg/m^2 Nanoparticle Paclitaxel | 45 mg/m^2 Nanoparticle Paclitaxel
Started | 3 (Includes participants from Phase I who were followed for efficacy but not retreated in Phase II.) | 51 (Includes participants from Phase I who were followed for efficacy but not retreated in Phase II.) | 3 (Includes participants from Phase I who were followed for efficacy but not retreated in Phase II.) | 55 (Includes participants from Phase I who were followed for efficacy but not retreated in Phase II.)
Completed | 3 | 49 | 3 | 50
Not Completed | 0 | 2 | 0 | 5
Not completed — Adverse Event | 0 | 2 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10 mg/m^2 Nanoparticle Paclitaxel | 22 mg/m^2 Nanoparticle Paclitaxel | 35 mg/m^2 Nanoparticle Paclitaxel | 45 mg/m^2 Nanoparticle Paclitaxel | Total
Number analyzed (Participants) | 3 | 51 | 3 | 55 | 112
Age Continuous [Mean (Standard Deviation); unit: years] | 63.7 (6.51) | 59.0 (9.26) | 63.3 (6.81) | 60.3 (8.89) | 59.9 (8.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 20 | 1 | 15 | 37
  Male | 2 | 31 | 2 | 40 | 75
Race/Ethnicity, Customized [Number; unit: participants]
  Black, of African Heritage | 0 | 1 | 0 | 3 | 4
  White, Non-Hispanic and Non-Latino | 3 | 44 | 3 | 46 | 96
  White, Hispanic or Latino | 0 | 6 | 0 | 6 | 12
Weight [Mean (Standard Deviation); unit: kg] | 82.80 (10.318) | 83.56 (13.659) | 91.33 (21.333) | 85.01 (17.915) | 84.46 (15.880)
Lesion type [Number; unit: participants]
  Patients with de novo Lesions | 3 | 49 | 3 | 50 | 105
  Patients with In-Stent Restenosis Lesions | 0 | 2 | 0 | 5 | 7
Diabetes mellitis [Number; unit: participants]
  No Diabetes | 3 | 40 | 2 | 46 | 91
  Insulin Dependent | 0 | 5 | 0 | 1 | 6
  Non-Insulin Dependent | 0 | 6 | 1 | 8 | 15
Minimum Lumen Diameter [Mean (Standard Deviation); unit: mm] — Participant population = 3, 47, 3, 50 (103 total). Measures were obtained from the angiographic evaluation.
  mm | 0.790 (0.3941) | 0.842 (0.3628) | 0.762 (0.1804) | 0.986 (0.3740) | 0.908 (0.3691)
Reference Diameter [Mean (Standard Deviation); unit: mm] — Participant population = 3, 50, 3, 54 (110 total). Measures were obtained from the angiographic evaluation.
  mm | 2.668 (0.0753) | 2.577 (0.3899) | 2.650 (0.4290) | 2.703 (0.4664) | 2.643 (0.4259)
Lesion Length [Mean (Standard Deviation); unit: mm] — Participant population = 3, 50, 3, 54 (110 total). Measures were obtained from the angiographic evaluation.
  mm | 6.342 (0.9086) | 10.720 (5.9338) | 7.900 (1.2630) | 10.067 (5.7097) | 10.203 (5.6932)
Diameter Stenosis [Mean (Standard Deviation); unit: % diameter stenosis] — Participant population = 3, 51, 3, 54 (111 total). Measures were obtained from the angiographic evaluation.
  % diameter stenosis | 80.92 (9.521) | 68.94 (15.083) | 70.50 (8.789) | 66.28 (14.253) | 68.01 (14.523)

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Number of Participants With Dose-limiting Toxicities
Description: Toxicities were evaluated based on the U.S. National Cancer Institute (NCI) Common Terminology Criteria (CTC) for Adverse Events version 3.0. Any drug-related toxicities considered CTC Grade 3 or 4 were considered dose limiting.
  The maximum tolerated dose was defined as the lesser of 45 mg/m^2 or the dose at which any drug related toxicities were observed.
Time Frame: Up to 1 week following percutaneous coronary intervention.
Population: Phase I treated population.
Measure: Number; unit: participants
Arm/Group | 10 mg/m^2 Nanoparticle Paclitaxel | 22 mg/m^2 Nanoparticle Paclitaxel | 35 mg/m^2 Nanoparticle Paclitaxel | 45 mg/m^2 Nanoparticle Paclitaxel
Number analyzed (Participants) | 3 | 3 | 3 | 3
participants | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Procedural Complications
Description: Procedural complications include the following:
  1. Haemodynamic monitoring: changes in heart rate, arterial blood pressure or electrocardiogram changes;
  2. Arrhythmia: premature ventricular complexes, brady or tachyarrhythmia;
  3. Allergic reactions: rash, flushing, pyrexia, urticaria, angio-oedema;
  4. Angiographic complications: coronary artery spasm, dissection, thrombosis, TIMI (Thrombolysis In Myocardial Infarction) flow, no reflow;
  5. Clinical changes: chest pain.
Time Frame: From Day 0 - Day 1 (from study drug administration until 24 hours post-procedure).
Population: Treated population.
Measure: Number; unit: participants
Arm/Group | 10 mg/m^2 Nanoparticle Paclitaxel | 22 mg/m^2 Nanoparticle Paclitaxel | 35 mg/m^2 Nanoparticle Paclitaxel | 45 mg/m^2 Nanoparticle Paclitaxel
Number analyzed (Participants) | 3 | 51 | 3 | 55
participants | 1 | 5 | 1 | 9
Statistical Analysis 1: Comparison: 22 mg/m^2 Nanoparticle Paclitaxel vs 45 mg/m^2 Nanoparticle Paclitaxel; The statistical testing of treatment difference is for exploratory purposes; Test type: Superiority or Other; p = 0.396, Fisher Exact

3. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs)
Description: An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.
  An SAE is any event that:
  * is fatal or life threatening
  * results in persistent or significant disability or or incapacity;
  * requires or prolongs existing hospitalization;
  * is a congenital anomaly/birth defect in the offspring of a patient who received medication;
  * conditions not included above that may jeopardize the patient or require intervention to prevent one of the outcomes listed above.
Time Frame: Up to 6 months.
Population: Treated population.
Measure: Number; unit: participants
Arm/Group | 10 mg/m^2 Nanoparticle Paclitaxel | 22 mg/m^2 Nanoparticle Paclitaxel | 35 mg/m^2 Nanoparticle Paclitaxel | 45 mg/m^2 Nanoparticle Paclitaxel
Number analyzed (Participants) | 3 | 51 | 3 | 55
participants
  Patients with at Least 1 AE | 3 | 43 | 3 | 48
  Patients with at Least 1 Serious AE | 0 | 14 | 0 | 18
Statistical Analysis 1: Comparison: 22 mg/m^2 Nanoparticle Paclitaxel vs 45 mg/m^2 Nanoparticle Paclitaxel; Comparison of the number of patients with any treatment emergent adverse event. The statistical testing of treatment difference is for exploratory purposes; Test type: Superiority or Other; p = 0.783, Fisher Exact

4. Secondary Outcome: Percentage of Participants With Binary Restenosis
Description: Binary restenosis was assessed by quantitative coronary angiography and defined as >50% diameter stenosis within the stented region (In-stent) or the stented region plus 5 mm on either side of the stent (In-segment) at follow-up. Angiograms were centrally assessed by the Angiographic Core Laboratory.
Time Frame: 6 months
Population: Treated Population.
Measure: Number; unit: percentage of participants
Arm/Group | 10 mg/m^2 Nanoparticle Paclitaxel | 22 mg/m^2 Nanoparticle Paclitaxel | 35 mg/m^2 Nanoparticle Paclitaxel | 45 mg/m^2 Nanoparticle Paclitaxel
Number analyzed (Participants) | 3 | 51 | 3 | 55
percentage of participants
  In-stent | 0.0 | 25.5 | 0.0 | 34.5
  In-segment | 0.0 | 27.5 | 0.0 | 34.5
Statistical Analysis 1: Comparison: 22 mg/m^2 Nanoparticle Paclitaxel vs 45 mg/m^2 Nanoparticle Paclitaxel; Comparison of in-stent binary restenosis. The statistical testing of treatment difference is for exploratory purposes; Test type: Superiority or Other; p = 0.293, Fisher Exact
Statistical Analysis 2: Comparison: 22 mg/m^2 Nanoparticle Paclitaxel vs 45 mg/m^2 Nanoparticle Paclitaxel; Comparison of in-segment binary restenosis. The statistical testing of treatment difference is for exploratory purposes; Test type: Superiority or Other; p = 0.400, Fisher Exact

5. Primary Outcome: Number of Participants With Major Adverse Cardiac Events (MACE) at 1 Month
Description: Major Adverse Cardiac Events (MACE) includes cardiac death, Coronary Artery Bypass Surgery, Myocardial Infarction, Target Vessel Revascularization (TVR) or Target Lesion Revascularization (TLR) and stent/vessel thrombotic occlusion.
Time Frame: From the day of Percutaneous Coronary Intervention to 1 Month.
Population: Treated population.
Measure: Number; unit: participants
Arm/Group | 10 mg/m^2 Nanoparticle Paclitaxel | 22 mg/m^2 Nanoparticle Paclitaxel | 35 mg/m^2 Nanoparticle Paclitaxel | 45 mg/m^2 Nanoparticle Paclitaxel
Number analyzed (Participants) | 3 | 51 | 3 | 55
participants | 0 | 1 | 0 | 1
Statistical Analysis 1: Comparison: 22 mg/m^2 Nanoparticle Paclitaxel vs 45 mg/m^2 Nanoparticle Paclitaxel; The statistical testing of treatment difference is for exploratory purposes; Test type: Superiority or Other; p > 0.999, Fisher Exact

6. Primary Outcome: Number of Participants With Major Adverse Cardiac Events (MACE) at 6 Months
Description: as for outcome 5
Time Frame: From the day of Percutaneous Coronary Intervention to Month 6.
Population: Treated population.
Measure: Number; unit: participants
Arm/Group | 10 mg/m^2 Nanoparticle Paclitaxel | 22 mg/m^2 Nanoparticle Paclitaxel | 35 mg/m^2 Nanoparticle Paclitaxel | 45 mg/m^2 Nanoparticle Paclitaxel
Number analyzed (Participants) | 3 | 51 | 3 | 54
participants | 0 | 7 | 0 | 16
Statistical Analysis 1: Comparison: 22 mg/m^2 Nanoparticle Paclitaxel vs 45 mg/m^2 Nanoparticle Paclitaxel; The statistical testing of treatment difference is for exploratory purposes; Test type: Superiority or Other; p = 0.061, Fisher Exact

7. Secondary Outcome: Late Lumen Loss
Description: Late lumen loss represents the extent of neointimal hyperplasia within the stented region (In-stent) or the stented region plus 5 mm on either side of the stent (In-segment) and was measured by quantitative coronary angiography.
  Late Loss = Minimum Lumen Diameter (MLD) Post Procedure minus the MLD at Follow-up.
Time Frame: Day 0 (post-procedure baseline) and 6 months.
Population: Treated population for whom data was available (indicated by "n").
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 10 mg/m^2 Nanoparticle Paclitaxel | 22 mg/m^2 Nanoparticle Paclitaxel | 35 mg/m^2 Nanoparticle Paclitaxel | 45 mg/m^2 Nanoparticle Paclitaxel
Number analyzed (Participants) | 3 | 51 | 3 | 55
mm
  In-stent [n=3, 46, 3, 50] | 0.403 (0.2267) | 0.871 (0.4188) | 0.747 (0.1626) | 0.835 (0.5328)
  In-segment [n=3, 47, 3, 50] | 0.281 (0.2116) | 0.631 (0.4070) | 0.355 (0.3101) | 0.697 (0.5323)
Statistical Analysis 1: Comparison: 22 mg/m^2 Nanoparticle Paclitaxel vs 45 mg/m^2 Nanoparticle Paclitaxel; Comparison of in-stent late lumen loss. The statistical testing of treatment difference is for exploratory purposes; Test type: Superiority or Other; p = 0.709, Fisher Exact
Statistical Analysis 2: Comparison: 22 mg/m^2 Nanoparticle Paclitaxel vs 45 mg/m^2 Nanoparticle Paclitaxel; Comparison of in-segment late lumen loss. The statistical testing of treatment difference is for exploratory purposes; Test type: Superiority or Other; p = 0.495, Fisher Exact

8. Secondary Outcome: Percentage of In-Stent Volume Obstruction at 6 Months
Description: In-stent volume obstruction at 6 months was measured by intra-vascular ultrasound (IVUS) and centrally assessed by the IVUS Core Laboratory. Percent in-stent volume obstruction was calculated as neointimal volume / stent volume * 100.
Time Frame: 6 months
Population: Treated population for whom data was available.
Measure: Mean (Standard Deviation); unit: Percentage of obstruction
Arm/Group | 10 mg/m^2 Nanoparticle Paclitaxel | 22 mg/m^2 Nanoparticle Paclitaxel | 35 mg/m^2 Nanoparticle Paclitaxel | 45 mg/m^2 Nanoparticle Paclitaxel
Number analyzed (Participants) | 3 | 40 | 3 | 43
Percentage of obstruction | 14.080 (11.5163) | 24.908 (15.3220) | 31.016 (8.9722) | 21.663 (14.0249)
Statistical Analysis 1: Comparison: 22 mg/m^2 Nanoparticle Paclitaxel vs 45 mg/m^2 Nanoparticle Paclitaxel; Test type: Superiority or Other; p = 0.317, ANOVA; P-value testing dose group differences based on an analysis of variance with dose effect in the model

ADVERSE EVENTS:
Time Frame: Up to 6 months.
Arm/Group | 10 mg/m^2 Nanoparticle Paclitaxel | 22 mg/m^2 Nanoparticle Paclitaxel | 35 mg/m^2 Nanoparticle Paclitaxel | 45 mg/m^2 Nanoparticle Paclitaxel
Serious Adverse Events (participants affected / at risk) | 0/3 | 14/51 | 0/3 | 18/55
Other Adverse Events (participants affected / at risk) | 3/3 | 34/51 | 3/3 | 31/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 10 mg/m^2 Nanoparticle Paclitaxel (N=3) | 22 mg/m^2 Nanoparticle Paclitaxel (N=51) | 35 mg/m^2 Nanoparticle Paclitaxel (N=3) | 45 mg/m^2 Nanoparticle Paclitaxel (N=55)
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 4 | 0 | 8
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 7
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 0 | 1
Chest discomfort (General disorders) | 0 | 1 | 0 | 0
Arterial disorder (Vascular disorders) | 0 | 1 | 0 | 0
Arterial restenosis (Vascular disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Coronary angioplasty (Surgical and medical procedures) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 10 mg/m^2 Nanoparticle Paclitaxel (N=3) | 22 mg/m^2 Nanoparticle Paclitaxel (N=51) | 35 mg/m^2 Nanoparticle Paclitaxel (N=3) | 45 mg/m^2 Nanoparticle Paclitaxel (N=55)
Aspartate aminotransferase increased (Investigations) | 2 | 4 | 1 | 3
Blood creatine phosphokinase MB increased (Investigations) | 2 | 4 | 0 | 3
Troponin T increased (Investigations) | 2 | 1 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 1
Electrocardiogram ST-T change (Investigations) | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 4 | 1 | 2
Troponin increased (Investigations) | 0 | 2 | 1 | 1
Chest discomfort (General disorders) | 1 | 1 | 0 | 0
Chest pain (General disorders) | 1 | 5 | 0 | 4
Pyrexia (General disorders) | 1 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 4 | 0 | 1
Oedema peripheral (General disorders) | 0 | 2 | 1 | 3
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 2
Paraesthesia (Nervous system disorders) | 1 | 2 | 0 | 0
Headache (Nervous system disorders) | 0 | 4 | 0 | 2
Presyncope (Nervous system disorders) | 0 | 3 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 1
Haematoma (Vascular disorders) | 1 | 4 | 1 | 3
Hypotension (Vascular disorders) | 0 | 4 | 0 | 5
Angina pectoris (Cardiac disorders) | 0 | 4 | 0 | 5
Contusion (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 5 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
* Study data will not be published in part before the complete multicenter data has been reported in full, unless more than 1 year has elapsed since completion of the Study.
* Investigator/institution must supply copy of presentation or publication to Celgene within 30 days of publication. Celgene may request in writing within that 30 days that Celgene Confidential Information be deleted or be granted a 60 day delay prior to publication to permit intellectual property filings.